CLINICAL TRIAL: NCT00460070
Title: Levetiracetam, Carbamazepine and Lamotrigine and Hormonal Side Effects in Adult Males and Females.
Brief Title: Study of Hormonal Sideeffects in Patients Taking Levetiracetam, Carbamazepine or Lamotrigine for Epilepsy
Status: Completed | Type: Observational
Sponsor: Rikshospitalet University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Erik Taubøll, Professor, Dep of Neurology, Rikshospitalet, OSLO
Other Study IDs: M52332
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2009-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Some antiepileptic drugs are found to have hormonal side effects. We want to study possible hormonal side effects of the relatively new antiepileptic drug; levetiracetam and compare it to the older drugs; lamotrigine and carbamazepine. The participants are going to fill in a questionnaire and we will collect blood samples from them, to analyse hormones.

DETAILED DESCRIPTION:
We have previously performed long-term studies of rats treated with levetiracetam and compared them with a control group. Here we have found that levetiracetam has a probable effect on the ovaries, since the treated animals had larger ovaries, fewer cysts, more corpora lutea and more secondary follicles than the untreated animals (Taubøll et al 2004). Blood tests on the animals showed that those treated with levetiracetam had higher testosterone levels and lower levels of estrogen and FSH, whilst LH and progesterone levels were unaffected by the treatment (Svalheim et al, 2005a, b). Studies on cell cultures from pig ovaries, as carried out by our group in collaboration with Jagiellonian University, Krakow, Poland, appeared to support these findings (Taubøll et al. 2006, submitted).

Our wish therefore now is to study fertile men and women in order to look for any changes in the balance of sex hormones during use of levetiracetam in order to establish whether the findings in animal trials are clinically relevant to humans.

ELIGIBILITY:
Inclusion Criteria:

* Having epilepsy
* Age 18- 45
* Using levetiracetam/ lamotrigine or carbamazepine in monotherapy for at least 6 months

Exclusion Criteria:

* Hormonal diseases( ie; diabetes, hypo/ hyperthyroid disease)
* Use of hormonal anticonception drugs or other hormonal drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from the outpatients clinic
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2007-01; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Taubøll, MD, Principal Investigator — unaffiliation
Locations (1):
- Dep. of Neurology, Rikshospitalet Universty Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Bachmann T, Bertheussen KH, Svalheim S, Rauchenzauner M, Luef G, Gjerstad L, Tauboll E. Haematological side effects of antiepileptic drug treatment in patients with epilepsy. Acta Neurol Scand Suppl. 2011;(191):23-7. doi: 10.1111/j.1600-0404.2011.01539.x. PMID 21711253
- [Result] Svalheim S, Luef G, Rauchenzauner M, Morkrid L, Gjerstad L, Tauboll E. Cardiovascular risk factors in epilepsy patients taking levetiracetam, carbamazepine or lamotrigine. Acta Neurol Scand Suppl. 2010;(190):30-3. doi: 10.1111/j.1600-0404.2010.01372.x. PMID 20586732
- [Result] Svalheim S, Tauboll E, Luef G, Lossius A, Rauchenzauner M, Sandvand F, Bertelsen M, Morkrid L, Gjerstad L. Differential effects of levetiracetam, carbamazepine, and lamotrigine on reproductive endocrine function in adults. Epilepsy Behav. 2009 Oct;16(2):281-7. doi: 10.1016/j.yebeh.2009.07.033. Epub 2009 Aug 27. PMID 19716343